CLINICAL TRIAL: NCT05614934
Title: Vonoprazan-based Therapy Versus Standard Regimen for Helicobacter Pylori Infection Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yumna Mohamed Shekeban, Teaching Assistant at clinical pharmacy and pharmacy practice department, faculty of pharmacy Alexandria University, Alexandria University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107175
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2022-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; vonoprazan; standard triple therapy

STUDY DESIGN:
Intervention Model Description: Open-labeled, prospective, three-arm, parallel-group, non-placebo Randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- S3 (Active Comparator): Standard clarithromycin triple
  Interventions: Drug: standard Clarithromycin triple therapy
- V3 (Experimental): Vonoprazan triple
  Interventions: Drug: Vonoprazan triple therapy
- V2 (Experimental): Vonoprazan dual
  Interventions: Drug: Vonoprazan dual therapy

INTERVENTIONS:
Drug: standard Clarithromycin triple therapy — Oral administration of proton pump inhibitor standard or double dose twice daily, clarithromycin 500 mg twice daily and, Amoxicillin1g twice daily for 14 days
  Arms: S3
Drug: Vonoprazan triple therapy — Oral administration of Vonoprazan 20mg twice daily, clarithromycin 500 mg twice daily, and, Amoxicillin1g twice daily for 14 days
  Arms: V3
Drug: Vonoprazan dual therapy — Oral administration of Vonoprazan 20mg twice daily and, Amoxicillin1g three times daily for 14 days
  Arms: V2

SUMMARY:
Appropriately, half of the global population is infected with H. pylori, and it is now recognized that it causes at least 95% of all gastric cancers. Currently, the main challenge in the field of H. pylori infection is the rapidly increasing antibiotic resistance worldwide, which is causing a decline in the effectiveness of currently available eradication regimens.

The aim of the study is to assess the safety and efficacy of different H. pylori vonoprazan-based regimens compared to the commonly used standard triple therapy composed of Clarithromycin, Amoxicillin, and Proton pump inhibitor to eradicate H. pylori infection in treatment-naive patients through the determination of each regimen eradication rate and reported safety profile

DETAILED DESCRIPTION:
1. Ethical committee approval is obtained from Ethics committee of Faculty of Medicine, Alexandria University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Patients with suspected H. pylori infection are recruited from Alexandria University out-patient clinics
4. Participants' demographic data, Full medical and medication history, and detailed clinical presentation is documented
5. Participants are tested for H. pylori infection using rapid H. pylori stool antigen test device
6. Negative subjects are excluded while positive patients are randomly allocated to 3 groups of different H. pylori regimens (Standard triple, Vonoprazan dual, and Vonoprazan triple)
7. Following up treatment side effects while taking the medications.
8. Assessing regimens effectiveness through patient retesting at least 1 month after treatment completion.
9. Assessing patient compliance to different regimens during the final visit.
10. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
11. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive stool antigen test result for H. pylori
* Patients recently diagnosed with H. pylori infection and did not receive any treatment

Exclusion Criteria:

* Patients sensitive to any of the regimens' components
* Patients who had received a previous eradication therapy and still show positive test results
* Recent use of antimicrobial agents, proton pump inhibitors, and H2 receptor blockers within 1 month
* Patients with gastric malignancy or who underwent previous gastric surgery
* Pregnancy and lactation
* Patients with major concomitant diseases, including psychic disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Determination of the eradication rates for each regimen | 1.5 month
  Percentage eradication in each group is calculated by intention-to-treat analysis or per-protocol analysis.

SECONDARY OUTCOMES:
Determination of number of compliant participants to each regimen | 1.5 month
  Adherence to therapies is determined through pill count in medication boxes In addition to reviewing a daily medication schedule filled by the participant.
Determination of number of participants with treatment related adverse events | 2 weeks
  Patients will be contacted on a regular basis to monitor any reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University outpatient clinics, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shekeban YM, Hamdy NA, Header DA, Ahmed SM, Helmy MM. Vonoprazan-based therapy versus standard regimen for Helicobacter pylori infection management in Egypt: an open-label randomized controlled trial. Sci Rep. 2025 May 8;15(1):15989. doi: 10.1038/s41598-025-98606-8. PMID 40341536